CLINICAL TRIAL: NCT03419364
Title: Phase II Study of Nicotinamide in Early Onset Preeclampsia
Brief Title: Study of Nicotinamide in Early Onset Preeclampsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0693; 1R03HD092370-01 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-07

CONDITIONS: Pre-Eclampsia; Pregnancy Related
MeSH Terms: conditions — Pre-Eclampsia | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: All participants will receive study agent. 2.5 gm nicotinamide given orally in 3 divided doses (1000 in morning, 500 in afternoon, 1000 at bedtime).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nicotinamide - pre-eclampsia (Experimental): All participants will receive study agent
  Interventions: Drug: nicotinamide
- Nicotinamide - healthy pregnant (Experimental): All participants will receive study agent 1000mg in single dose
  Interventions: Drug: nicotinamide
- Healthy Non-Pregnant (Experimental): All participants will receive study agent 1000mg in single dose
  Interventions: Drug: nicotinamide

INTERVENTIONS:
Drug: nicotinamide — 2.5 gm nicotinamide given orally in 3 divided doses: 1000 mg in morning and evening, 500 mg at noon/midday
  Other Names: niacinamide

SUMMARY:
Phase II Study of 2.5 gm of nicotinamide, given daily in 3 divided doses, to measure effect on maternal blood pressure in women with early onset preeclampsia and to determine peak and trough levels of nicotinamide. We will compare peak and trough levels in healthy non-pregnant and healthy pregnant participants.

DETAILED DESCRIPTION:
See brief summary above

ELIGIBILITY:
Diagnosis and Inclusion Criteria

* Maternal age 18-55 years
* Singleton pregnancy with no known fetal anomalies
* Early-onset preeclampsia OR early-onset severe gestational hypertension defined as:

  * Early-onset: between 24 weeks 0 days and -33 weeks 3 days, based on menstrual dating confirmed by first or second trimester ultrasound OR second trimester ultrasound if menstrual dating unavailable;
  * Preeclampsia:
* New onset hypertension and proteinuria, with systolic BP > 140 mm Hg and/or diastolic BP > 90 mm Hg on two occasions 6 hours apart and > 300 mg proteinuria on 24 hour urine collection OR urine P/C ratio >0.3;
* New onset hypertension and NO proteinuria, with systolic BP > 140 mm Hg and/or diastolic BP > 90 mm Hg on two occasions 6 hours apart and one or more of the following: serum creatinine >1.1 mg/dL or doubling from baseline ,or central nervous system symptoms or visual changes
* Severe preeclampsia defined as new onset systolic BP > 160 mm Hg and/or diastolic BP > 105 with proteinuria as above or or without proteinuria and one or more of the following criteria listed above

  * Candidate for expectant management for at least 48 hours
  * Deemed clinically stable by primary clinician and candidate for expectant management (delayed delivery) for at least 48 hours;
* Maternal liver function tests < 2x ULN
* Maternal platelet count > 100,000 mm³
* Planned expectant management
* Pre-existing medical diseases such as hypertension, diabetes, endocrine disorders, gastrointestinal diseases, are well controlled
* Fetal well-being established by estimated fetal weight > 5th %tile; normal amniotic fluid volume (MVP > 2 cm); normal Umbilical Artery (UA) Dopplers; or reactive Non Stress Test (NST) or Biophysical Profile (BPP) > 6
* Delivery not anticipated within 48 hours of enrollment

Exclusion Criteria

* Pre-existing renal disease (creatinine > 1.5 mg/dL)
* Any pre-existing medical condition that would increase risk for liver toxicity (e.g. hepatitis B or C; HIV; Isoniazid (INH) use)
* Eclampsia; cerebral edema on CT/MRI; headache unrelieved by analgesics
* Evidence of liver dysfunction (LFTs > 2x ULN)
* Thrombocytopenia (platelets < 100,000 mm³)
* Pulmonary edema
* HELLP syndrome
* Evidence of fetal compromise: Estimated Fetal Weight (EFW) < 5th percentile; or BPP < 6; or absent or reverse diastolic UA blood flow; or oligohydramnios (MVP < 2 cm)
* Placental abruption defined as unexplained vaginal bleeding
* Preterm labor defined as regular contractions and cervical change
* Any condition deemed by the investigator to be a risk to mother or fetus in completion of the study
* Any condition deemed by the investigator to require delivery within 48 hours

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study of pregnant and non-pregnant women only
Enrollment: 23 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Boggess, MD, Principal Investigator — UNC_Chapel Hill
Locations (1):
- UNC at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotinamide - Healthy Pregnant; Nicotinamide - Healthy Non-Pregnant: All participants will receive study agent 1000 mg in single dose
  nicotinamide: 1000 mg nicotinamide in morning
Period: Overall Study
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Started | 11 | 6 | 6
Signed Consent | 11 | 6 | 6
Received Intervention | 9 | 6 | 6
Completed | 9 | 6 | 6
Not Completed | 2 | 0 | 0
Not completed — Delivery due to maternal condition | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant | Total
Number analyzed (Participants) | 9 | 6 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 6 | 21
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 6 | 21
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 6 | 6 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 4 | 6 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 6 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Arterial Blood Pressure (MAP)
Description: Blood pressure (mmHg) will be used to observe the effect of nicotinamide. The highest MAP (defined as the highest MAP within the 24 hour period prior to the administration of study agent) and the highest MAP through 24 hours after study drug administration.
Time Frame: Baseline, 48 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 6 | 6
mmHg | 0 (9) | 2 (9) | 4 (6)

2. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) =/> 3x Upper Limit of Normal (ULN)
Time Frame: Within 24 hours of any dose, up to a maximum 4 weeks
Population: Healthy women were not at risk for liver toxicity and therefore were not assessed for ALT.
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 0 | 0
Participants | 0 |  |

3. Secondary Outcome: Number of Participants With Aspartate Aminotransferase (AST) =/> 3x Upper Limit of Normal (ULN)
Time Frame: Within 24 hours of any dose, up to a maximum 4 weeks
Population: Healthy women were not at risk for liver toxicity and therefore were not assessed for AST.
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 0 | 0
Participants | 0 |  |

4. Secondary Outcome: Number of Participants With Maternal Side Effects
Description: Maternal side effects are defined as: facial erythema, hives, sore mouth, dry hair, fatigue, flushing, headache, nausea, and heart burn.
Time Frame: From initial administration of study agent until 24 hours post last dose, up to a maximum of 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 6 | 6
Participants | 0 | 0 | 0

5. Secondary Outcome: Percentage of Women Maternal Abdominal Tenderness
Time Frame: From initial administration of study agent until 24 hours post last dose, up to a maximum of 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 6 | 6
percentage of participants | 0 | 0 | 0

6. Secondary Outcome: Percentage of Women With Headache Unrelieved by Oral Analgesics
Time Frame: From initial administration of study agent until 24 hours post last dose, up to a maximum of 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 6 | 6
percentage of participants | 33 | 0 | 0

7. Secondary Outcome: Percentage of Women With Hematocrit Decrease of More Than 3%
Time Frame: From initial administration of study agent until 24 hours post last dose, up to a maximum of 4 weeks
Population: Healthy women were not at risk for anemia and therefore were not assessed for Hematocrit.
Measure: Number; unit: percentage of participants
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 0 | 0
percentage of participants | 44 |  |

8. Secondary Outcome: Percentage of Women With Less Than 500 cc Urine Output in 24 Hours
Time Frame: From initial administration of study agent until 24 hours post last dose, up to a maximum of 4 weeks
Population: Healthy women were not at risk for oliguria and therefore were not assessed for urine output.
Measure: Number; unit: percentage of participants
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 0 | 0
percentage of participants | 0 |  |

9. Secondary Outcome: Percentage of Fetuses With Category III Non Stress Test Results
Description: A Non Stress Test is a determination of the current well-being of the fetus, as measured by the fetal heart rate. Category I indicates that the fetus is in a state of well-being and is tolerating the intrauterine environment. Category II indicates a fetal heart rate that is showing some signs of distress. In this instance, obstetric providers will try to improve the intrauterine environment to allow the pregnancy to continue. Category III relates to a fetus whose well-being is compromised - usually requiring rapid intervention, ie expedient delivery.
Time Frame: From initial administration of study agent until 24 hours post last dose, up to a maximum of 4 weeks
Population: Healthy women were not at risk for placental insufficiency and therefore did not have a non stress test.
Measure: Number; unit: percentage of fetuses
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 9 | 0 | 0
percentage of fetuses | 0 |  |

10. Secondary Outcome: Percentage of Fetuses With Biophysical Profile < 6
Time Frame: From initial administration of study agent until 24 hours post last dose
Population: Data only collected if indicated and performed as part of clinical care. No primary care providers felt this test was indicated.
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Mean Peak Nicotinamide Level
Description: The mean was calculated for each group using blood samples drawn on Day 1 at 1 hour post 1000 mg nicotinamide administration routinely given at 8 a.m. Peak nicotinamide level expected at 1 hour post dose.
Time Frame: at 1 hour post 1000 mg nicotinamide administration on Day 1
Population: Data reported for all participants who had blood collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 12701.7 (6187.5) | 13279.7 (970.7) | 16314.1 (3337.1)

12. Secondary Outcome: Mean Trough Concentration Nicotinamide Administration
Description: The mean was calculated for each group for blood samples drawn on Day 1 8 hours post 1000 mg nicotinamide administration routinely given at 8 a.m. Trough nicotinamide level is measured immediately prior to the next dose.
Time Frame: 8 hours after the 8 a.m. 1000 mg nicotimamide administration on Day 1
Population: Data reported for all participants who had blood collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 479.2 (967.3) | 1490.7 (1907.8) | 1991.2 (2783.6)

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 30 days after infant delivery, ranging from 31 to 58 days total.
Arm/Group | Nicotinamide - Pre-eclampsia | Nicotinamide - Healthy Pregnant | Nicotinamide - Healthy Non-Pregnant
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03419364/Prot_SAP_000.pdf